CLINICAL TRIAL: NCT02012530
Title: A Cohort Comparison Study Comparing Platelet Rich Plasma vs Hyaluronic Acid Intra-articular Knee Injections for Early Cartilage Defects in the Knee
Brief Title: PRP vs HA Intra-articular Knee Injections for Cartilage Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shetty-Kim Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKRF 003
Record Dates: First submitted 2013-10-11; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis
Keywords: Articular cartilage; Hyaluronic Acid (HA); Platelet rich plasma (PRP)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HA (Active Comparator): Patients in this arm will have hyaluronic acid (HA) injected into their knee along with 3 ml local anaesthetic. The HA injection is in the form of 2 ml aqueous sodium hyaluronate. The exact constituents of the HA change in a proprietary manner. All HA injections used will have the CE marking on them.
  Interventions: Procedure: HA
- PRP (Active Comparator): Patients in this arm will have platelet rich plasma (PRP) injected into their knee. The PRP sample will be produced at the time of the injection. 30 ml of blood is drawn fro the patient a few minutes before the injection. Using a CE marked differential centrifugation device, the platelets are isolated. This concentrated sample of platelets is injected into the knee after the skin around the injection site is anaesthetised with local anaesthetic.
  Interventions: Procedure: PRP

INTERVENTIONS:
Procedure: HA — HA is widely applied in clinical practice with good results in many studies. HA forms part of the inflammatory process that can lead to the regeneration of cartilage in defective areas of the knee.
  Arms: HA
Procedure: PRP — PRP uses reparative growth factors taken from the patient's own blood to create an environment in the knee conducive to wound healing that can fill cartilage defects. It's autologous origin, easy preparation and safety profile makes it a potentially ground breaking treatment option for knee cartilage defects and osteoarthritis.
  Arms: PRP

SUMMARY:
Study Title: A cohort comparison study Comparing Platelet Rich Plasma vs Hyaluronic Acid Intra-articular Knee Injections for Early Cartilage Defects in the knee.

Study hypothesis: We start with the hypothesis that both treatments are equally effective.

Trial Design: The participating patients will be divided into two groups, each group receiving either one of the treatment modalities. This study will be randomised. Both procedures will be done at the Spire Alexandra Hospital by Professor A. A Shetty. The post-operative rehabilitation process will be the same for both groups.

Trial Participants: All participants will be from patients attending Professor Shetty's clinic at the Spire Alexandra Hospital.

Planned Sample Size: 50 patients in each group

Follow-up duration: The participating patients will be followed up at 2 weeks, 6 weeks, 3 months following the surgery by visits to the clinic and assessed clinically. The surgical outcomes will be measured by by IKDC, KOOS and Lysholm scores.

Planned Trial Period: Two to three years

Primary Objective: To establish superiority, if any, of either procedure over the other by studying pain relief, improvement in function.

Primary Endpoint: At the end of the 2 year follow up for all participating patients.

DETAILED DESCRIPTION:
Osteoarthritis and early degenerative cartilage lesions has a significant impact on our society. People are both living and are more active for longer and so their demands are greater. This is having a direct effect on our economy from days missed off work and greater dependency on state resources.

The limited regenerative capacity of cartilage is part of this problem. Existing degenerative lesions lead to accelerated deterioration of the articular (joint) surface leading to end-stage arthritis. Any solution that can delay or reverse this process is therefore desirable. A number of non-invasive solutions do exist to treat painful knees that improve functionality but with varying rates of success. Two of the more promising agents are hyaluronic acid (HA) and platelet rich plasma (PRP). HA is widely applied in clinical practice with good results in many studies. HA forms part of the inflammatory process that can lead to the regeneration of cartilage in defective areas of the knee.

PRP uses reparative growth factors taken from the patient's own blood to create an environment in the knee conducive to wound healing that can fill cartilage defects. It's autologous origin, easy preparation and safety profile makes it a potentially ground breaking treatment option for knee cartilage defects and osteoarthritis.

These solutions work to improve the localised environment of morbidity and so for this reason are best administered as intra-articularly. As PRP is still in the earlier stages of its development, its exact dosage is still to be determined. HA has also recently been prepared as a higher concentration solution to test if there are any benefits to this.

Trials have compared these two products. No randomised controlled trials exist making our proposed research important.

Our null hypothesis is that there is no difference between HA and PRP in treating patients will articular lesions.

We will attempt to answer our research question by means of a randomised trial as there have been no trials to date that have proposed to clarify this clinical question. The reason for choosing a randomised trial is that it will take the quality of our research findings to a higher level than already exists in the literature. PRP will be compared with HA as these are two products with similar objectives. HA has been used for longer and has a more proven clinically successful track record. Selected participants will be randomised to receive either HA or PRP intra-articular injections.

Patients will be sourced from GP referrals to our knee unit clinic at the Alexandra Spire Hospital. Post-arthroscopy patients or existing follow up patients that satisfy the inclusion criteria will also be offered a place in our trial. Selected patients will be given a participant information sheet to read that will explain all about the trial. They will meet an investigator (doctor) to answer any queries and sign a consent form if they so wish.

Upon inclusion they will fill out a scoring questionnaire, be randomised and receive their corresponding injection. PRP recipients will have a sample of blood taken as is the requirement for the procedure.

They will then be followed up in clinic at 6 weeks, 3, 6, and 12 months where they will have to fill in a scoring questionnaire each time. The trial will therefore last from inclusion of our first patient until the last patient is followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

Participant is willing and able to give informed consent for participation in the study.

* Male or Female, aged 18 years or above.
* Diagnosed with either early degenerative cartilage lesions (Grade 1-3) as determined by plain radiograph, MRI or intra-operatively (categorised as per Outerbridge/ICRS classification).
* The patient must have more than a four month history of knee pain or swelling whether continuous or intermittent.

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Systemic disorders- DM, RA, SLE
* Major axial deviation (varus>5˚, valgus>5˚)
* Patients suffering from haematological disorders (coagulopathy)
* Patients with severe cardiovascular disease
* Active infection
* Immuno-suppressed patients
* Patients taking anticoagulants such warfarin or low molecular weight heparin
* Haemoglobin levels below 11g/dl
* Platelet count below 150000/mmc
* Participants who have participated in another research study involving an investigational product in the past 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 3 months
  The participating patients will be followed up at 2 weeks, 6 weeks and finally at 3 months following the injection by visits to the clinic and assessed clinically. The surgical outcomes will be measured by by KOOS score.

SECONDARY OUTCOMES:
Change in VAS Score at 3 months | 3 months
  The Participants will be followed at at 2 weeks, 6 weeks and finally at 3 months following the injection and will be asked to score a Visual Analogue Scale for pain at every visit. These scores will be compared to pre-operative values.

CONTACTS AND LOCATIONS:
Overall Officials: Asode A Shetty, MD, MCh, PhD, FRCS, Principal Investigator — Canterbury Christ Church University
Locations (1):
- Kent Knee Unit, Walderslade, Kent, United Kingdom